CLINICAL TRIAL: NCT06836128
Title: The Combined Effect of N-Acetyl Cysteine and Metformin in Polycystic Ovary Syndrome Patients
Acronym: PCOS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Marwa Rafat Talat, Demonstrator and Teaching assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Acetylcysteine in PCOS
Record Dates: First submitted 2025-01-30; First posted 2025-02-20 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS; NAC; metformin
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, interventional, open-label controlled parallel design study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group-MN (Experimental): Group-MN, constituting 51 cases, will receive N-acetyl cysteine and metformin (600 mg three times daily of acetyl cysteine and 500 mg once daily for one week, then 500 mg twice daily for one week, and 500 mg three times daily thereafter of metformin)
  Interventions: Drug: N-acetyl cysteine; Drug: Metfomin
- Group-M (Experimental): Group-M, constituting 51 cases, will receive treatment with metformin (starting with 500 mg once daily for one week, then 500 mg twice daily for one week, and 500 mg three times daily thereafter)
  Interventions: Drug: Metfomin

INTERVENTIONS:
Drug: N-acetyl cysteine — N-Acetyl Cysteine (NAC) has antioxidant properties and is essential for the body's production of glutathione, and both glutathione and NAC are potent antioxidants.
  Other Names: NAC
  Arms: Group-MN
Drug: Metfomin — metformin is commonly used for managing polycystic ovary syndrome (PCOS) due to its benefits in addressing several underlying features of the condition. While it is not officially approved by regulatory agencies like the FDA for PCOS, it is widely recognized and recommended in clinical practice guidelines as an off-label treatment for PCOS, particularly in women with insulin resistance and metabolic dysfunction.

SUMMARY:
The study aims to evaluate the effects of combination of metformin with NAC in PCOS on biochemical and hormonal parameters.

DETAILED DESCRIPTION:
Polycystic ovarian syndrome (PCOS) is one of the prevalent endocrine illnesses that affects women in industrialized and developing nations, with a prevalence that ranges from 8% to 13%. The most widely accepted criteria for diagnosing polycystic ovary syndrome (PCOS) are the Rotterdam criteria established in 20032. According to these criteria, a diagnosis is made if a patient meets at least two of the following three criteria:

The Rotterdam criteria

Polycystic ovarian syndrome is diagnosed when 2 out of 3 criteria are met:

1. Oligo-or/and anovulation
2. Clinical hyperandrogenism (acne, hirsutism, alopecia) or biochemical hyperandrogenism.
3. Polycystic ovarian morphology on transvaginal ultrasonography or high antimullerian hormone.

And exclusion of other etiologies (congenital adrenal hyperplasia, androgen-secreting tumors, Cushing's syndrome).

The 2023 International Evidence-based Guideline for the Assessment and Management of PCOS has built on the Rotterdam criteria by emphasizing more comprehensive assessments.

These updates highlight the need to consider a broader range of phenotypes, assess metabolic risks, and prioritize patient-centered, individualized care.

Algorithm: Screening and diagnostic assessment

Step 1:

Irregular Menstrual Cycles + Clinical Hyperandrogenism

• Exclude other causes* = diagnosis.

Step 2:

Irregular Menstrual Cycles Without Clinical Hyperandrogenism • Test for biochemical hyperandrogenism and exclude other causes* = Diagnosis

Step 3:

If Only Irregular Cycles or Only Hyperandrogenism

1. Adolescents: Ultrasound or AMH is not indicated = considered at risk of PCOS and reassessed later
2. Adults: Ultrasound for Polycystic Ovarian morphology (PCOM)* OR Anti-Mullerian Hormone (AMH) level, if positive (exclude other causes) * = diagnosis

   * Exclusion of Other Causes = TSH, prolactin, FSH or, if clinically indicated, exclude other causes (e.g. Cushing's syndrome, adrenal tumors, etc.) Irregular menstrual cycles 1 to < 3 years post-menarche: Cycle length is either less than 21 days or more than 45 days.

> 3 years post-menarche until perimenopause: Cycle length is either less than 21 days, more than 35 days, or fewer than 8 cycles per year.

> 1-year post-menarche: Any cycle lasting more than 90 days. Primary amenorrhea: no menstruation by age 15 or more than 3 years after the onset of breast development (thelarche).

Biochemical hyperandrogenism Elevated total or free testosterone, or calculated indices of free testosterone Clinical hyperandrogenism Comprehensive history and physical examination are needed. Adults: acne, female pattern hair loss, and hirsutism. Adolescents: severe acne and hirsutism.

Note the negative psychosocial impact of clinical hyperandrogenism. Standardized visual scales are preferred, including the modified Ferriman Gallway score (mFG), a score of ≥ 4-6 = hirsutism.

Ultrasound and polycystic ovary morphology (PCOM) and anti-mullerian hormone (AMH) Using ultrasound transducers with a frequency bandwidth including 8 MHz, the PCOM threshold is a follicle number per ovary of ≥ 20 and/or an ovarian volume ≥ 10 ml on either ovary, avoiding corpora lutea, cysts or dominant follicles.

Either serum AMH OR ultrasound may be used but not both to avoid overdiagnosis Serum AMH could be used for defining PCOM in adults as an alternative to pelvic or abdominal ultrasound.

People with PCOS often experience various metabolic and reproductive outcomes such as obesity, insulin resistance (IR), oxidative stress (OS), hirsutism, acne, irregular menstruation, and infertility, as well as long-term consequences including cancer and cardiovascular illnesses.

The cause of PCOS is still unknown, despite evidence indicating the pathophysiology of the condition is primarily driven by the production of high quantities of androgen and IR. Additionally, research showed that OS is linked to IR, hyperinsulinemia, hyperandrogenism, persistent inflammatory conditions, abnormalities in fat and carbohydrate metabolism, ovarian dysfunction, and unfavorable pregnancy outcomes. Consequently, antioxidant therapy might be useful in the management of PCOS. Patients with PCOS frequently seek treatment for a variety of symptoms, including menstrual irregularities, heavy menstrual bleeding, acne, hirsutism, and weight management challenges.

The management of PCOS is typically tailored to address these specific symptoms, with a range of therapeutic options available depending on the patient's presentation. Menstrual irregularity and heavy bleeding in patients with PCOS can be managed through lifestyle interventions, such as diet and exercise aimed at achieving a weight reduction of 5%-10%8, or by using combined hormonal contraceptives. These may include oral norethindrone acetate (5 mg daily for 7 days every 30-90 days, or 5 mg daily for 3 weeks on and 1 week off), ethinyl estradiol (20-35 mcg of ethinyl estradiol in combination with a progestin), or oral drospirenone (4 mg for 24 days, followed by 4 days of placebo). In cases where hormonal contraceptives are not suitable or effective, metformin (1500-2000 mg daily in divided doses, starting at 500 mg and increasing by 500 mg every 1-2 weeks) may be considered. Inositol supplementation, commonly administered as 4 g of myo-inositol daily, is another option that has been shown to improve menstrual regularity, metabolic disturbances, and reducing weight in patients with PCOS.

For managing acne, hirsutism, or alopecia, first-line treatments include combined hormonal contraceptives to address androgenic symptoms. In addition, topical treatments for hirsutism, such as 13% eflornithine, can help reduce unwanted facial hair. Minoxidil (2% solution, applied twice daily) is commonly used for the treatment of alopecia. Topical or oral acne treatments should follow general dermatological guidelines, depending on the severity of the condition.

Overweight or obesity is commonly addressed through lifestyle interventions. Metformin (1500-2000 mg daily in divided doses, with gradual titration starting at 500 mg) can be used to improve insulin sensitivity and aid in weight management.

For ovulation induction, letrozole (2.5 mg-7.5 mg for 5 days) is considered a first-line treatment for ovulation induction in many guidelines. To confirm successful ovulation, it is recommended to measure serum progesterone levels approximately 3 weeks after initiating letrozole. Metformin (1500-2000 mg daily) can also be used to enhance ovulatory function. Clomiphene is also used to induce ovulation, starting at 50 mg daily for 5 days from days 2-5 of the cycle. If ineffective, the dose may be increased to 100 mg or 150 mg in subsequent cycles for up to 6 cycles.

N-Acetyl Cysteine (NAC) has antioxidant properties and is essential for the body's production of glutathione, and both glutathione and NAC are potent antioxidants. By promoting the synthesis of glutathione synthetase hormone (GSH), NAC helps inhibit OS, preventing hyperinsulinemia-induced IR and protecting insulin receptors from oxidative damage. NAC likely enhances insulin receptor activity, leading to increased glucose consumption, which indicates improved insulin sensitivity. IR, dyslipidemia, and hyperhomocysteinemia are risk factors for ischemic heart disease in women with PCOS. NAC has been utilized as a therapeutic agent to improve homocysteine levels and lipid profiles, which in turn have been shown to affect insulin receptor activity. As a result, the primary cause of PCOS was alleviated and insulin levels fell. The antioxidant properties of NAC have been utilized in multiple clinical trials conducted on infertile PCOS females to increase oocyte quality and ovulation rate.

In this study, the investigators will evaluate and compare the efficacy of metformin and NAC combination versus metformin alone on clinical, metabolic, hormonal, and biochemical aspects in patients with PCOS.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged 20 to 45 years old.
2. Confirmed diagnosis with PCOS according to the 2023 International Evidence-based Guideline for the Assessment and Management of PCOS.
3. Ability to give informed consent.

Exclusion Criteria:

1. Hypersensitivity to either metformin or NAC.
2. Consumption of medications affecting carbohydrate metabolism, such as insulin, sulfonylureas, and taking hormonal analogues two months prior to enrollment.
3. Hyperprolactinemia, defined as a prolactin level above laboratory reference range.
4. Diabetes mellitus.
5. Thyroid dysfunction, subjects with elevated or low TSH level.
6. Renal impairment where creatinine clearance (CrCl) less than 30 ml/min.
7. Severe hepatic impairment, defined as significant biochemical abnormalities, including hypoalbuminemia and abnormal serum concentration (2-3 times the upper limit of normal), of at least two of the following liver function markers: total bilirubin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), or gamma-glutamyl transferase (GGT).
8. Active alcohol abuse.
9. History of lactic acidosis during metformin therapy.
10. Active peptic ulcer.
11. Congenital adrenal hyperplasia.
12. Cushing's syndrome.
13. Androgen secreting neoplasia.
14. Patients who were using spironolactone, other anti-androgens, or any form of hormone therapy for the treatment of hirsutism at least 3 months before enrollment in the study.
15. Decompensated heart failure.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 102 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcome will be change in LH/FSH levels. | 3 months
  change in LH/FSH ratio

SECONDARY OUTCOMES:
improvement in hormonal levels in patients with PCOS | 3 months
  Hormonal profile change in:
  Total testosterone levels (ng/dL) Free testosterone levels (ng/dL) Free testosterone to total testosterone (FT/TT) ratio, calculated from the measured values.
improvement in clinical features in patients with PCOS | 3 months
  improvement in clinical features: Menstrual irregularities: improvement in oligomenorrhea or amenorrhea, assessed based on The 2023 International Evidence-based Guideline for the Assessment and Management of PCOS Hirsutism: Assessed using the modified Ferriman-Gallwey (mFG) score Acne: Evaluated using the Investigator Global Assessment (IGA) scale technique.
improvement in biochemical parameters in patients with PCOS | 3 months
  biochemical parameters change in: Fasting insulin levels (µIU/mL). Fasting blood glucose (FBG) levels (mg/dL). Glucose/insulin ratio, calculated using fasting glucose and insulin levels. Homeostatic Model Assessment of Insulin Resistance (HOMA-IR), calculated using the standard formula.
improvement in metabolic parameters in patients with PCOS | 3 months
  weight in kilograms, height in meters Body mass index (BMI) (kg/m2), calculated as weight (kg) divided by height (m2).

CONTACTS AND LOCATIONS:
Overall Officials: Samar F Farid, PhD, Study Director — Professor and Head of Clinical Pharmacy Department, Faculty of Pharmacy, Cairo University; Eglal A Mostafa Bassiouny, PhD, Study Director — Lecturer of Clinical Pharmacy Faculty of Pharmacy, Cairo University; Amr Z Abdelhamid, PhD, Study Director — Obstetrics and Gynaecology Lecturer Kasr Al-Ainy School of Medicine, Cairo University
Locations (1):
- Kasr El-Ainy hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tiganis T. Reactive oxygen species and insulin resistance: the good, the bad and the ugly. Trends Pharmacol Sci. 2011 Feb;32(2):82-9. doi: 10.1016/j.tips.2010.11.006. Epub 2010 Dec 14. PMID 21159388
- [Background] Pei Y, Liu H, Yang Y, Yang Y, Jiao Y, Tay FR, Chen J. Biological Activities and Potential Oral Applications of N-Acetylcysteine: Progress and Prospects. Oxid Med Cell Longev. 2018 Apr 22;2018:2835787. doi: 10.1155/2018/2835787. eCollection 2018. PMID 29849877
- [Background] Yifu P. A review of antioxidant N-acetylcysteine in addressing polycystic ovary syndrome. Gynecol Endocrinol. 2024 Dec;40(1):2381498. doi: 10.1080/09513590.2024.2381498. Epub 2024 Jul 22. PMID 39039898
- [Background] Christ JP, Cedars MI. Current Guidelines for Diagnosing PCOS. Diagnostics (Basel). 2023 Mar 15;13(6):1113. doi: 10.3390/diagnostics13061113. PMID 36980421
- [Background] Gayatri K, Kumar JS, and Kumar BB. Metformin and N-acetyl cysteine in polycystic ovarian syndrome--a comparative study. Indian Journal of Clinical Medicine. 2023;15;24(18):14126. doi.org/10.1177/117739361000100002
- [Background] Scholze A, Rinder C, Beige J, Riezler R, Zidek W, Tepel M. Acetylcysteine reduces plasma homocysteine concentration and improves pulse pressure and endothelial function in patients with end-stage renal failure. Circulation. 2004 Jan 27;109(3):369-74. doi: 10.1161/01.CIR.0000109492.65802.AD. Epub 2004 Jan 19. PMID 14732754
- [Background] Fulghesu AM, Ciampelli M, Muzj G, Belosi C, Selvaggi L, Ayala GF, Lanzone A. N-acetyl-cysteine treatment improves insulin sensitivity in women with polycystic ovary syndrome. Fertil Steril. 2002 Jun;77(6):1128-35. doi: 10.1016/s0015-0282(02)03133-3. PMID 12057717
- [Background] De Mattia G, Bravi MC, Laurenti O, Cassone-Faldetta M, Proietti A, De Luca O, Armiento A, Ferri C. Reduction of oxidative stress by oral N-acetyl-L-cysteine treatment decreases plasma soluble vascular cell adhesion molecule-1 concentrations in non-obese, non-dyslipidaemic, normotensive, patients with non-insulin-dependent diabetes. Diabetologia. 1998 Nov;41(11):1392-6. doi: 10.1007/s001250051082. PMID 9833950
- [Background] Brown J, Farquhar C. Clomiphene and other antioestrogens for ovulation induction in polycystic ovarian syndrome. Cochrane Database Syst Rev. 2016 Dec 15;12(12):CD002249. doi: 10.1002/14651858.CD002249.pub5. PMID 27976369
- [Background] Costello M, Garad R, Hart R, Homer H, Johnson L, Jordan C, Mocanu E, Qiao J, Rombauts L, Teede HJ, Vanky E, Venetis C, Ledger W. A Review of First Line Infertility Treatments and Supporting Evidence in Women with Polycystic Ovary Syndrome. Med Sci (Basel). 2019 Sep 10;7(9):95. doi: 10.3390/medsci7090095. PMID 31510088
- [Background] Martin KA, Anderson RR, Chang RJ, Ehrmann DA, Lobo RA, Murad MH, Pugeat MM, Rosenfield RL. Evaluation and Treatment of Hirsutism in Premenopausal Women: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2018 Apr 1;103(4):1233-1257. doi: 10.1210/jc.2018-00241. PMID 29522147
- [Background] Greff D, Juhasz AE, Vancsa S, Varadi A, Sipos Z, Szinte J, Park S, Hegyi P, Nyirady P, Acs N, Varbiro S, Horvath EM. Inositol is an effective and safe treatment in polycystic ovary syndrome: a systematic review and meta-analysis of randomized controlled trials. Reprod Biol Endocrinol. 2023 Jan 26;21(1):10. doi: 10.1186/s12958-023-01055-z. PMID 36703143
- [Background] Teede HJ, Misso ML, Costello MF, Dokras A, Laven J, Moran L, Piltonen T, Norman RJ; International PCOS Network. Recommendations from the international evidence-based guideline for the assessment and management of polycystic ovary syndrome. Fertil Steril. 2018 Aug;110(3):364-379. doi: 10.1016/j.fertnstert.2018.05.004. Epub 2018 Jul 19. PMID 30033227
- [Background] Dason ES, Koshkina O, Chan C, Sobel M. Diagnosis and management of polycystic ovarian syndrome. CMAJ. 2024 Jan 28;196(3):E85-E94. doi: 10.1503/cmaj.231251. No abstract available. PMID 38286488
- [Background] Schuring AN, Schulte N, Sonntag B, Kiesel L. Androgens and insulin--two key players in polycystic ovary syndrome. Recent concepts in the pathophysiology and genetics of polycystic ovary syndrome. Gynakol Geburtshilfliche Rundsch. 2008;48(1):9-15. doi: 10.1159/000111465. Epub 2008 Jan 17. PMID 18209494
- [Background] Zeber-Lubecka N, Ciebiera M, Hennig EE. Polycystic Ovary Syndrome and Oxidative Stress-From Bench to Bedside. Int J Mol Sci. 2023 Sep 15;24(18):14126. doi: 10.3390/ijms241814126. PMID 37762427
- [Background] International Evidence-Based Guideline for the Assessment. 2023, www.monash.edu/__data/assets/pdf_file/0003/3379521/Evidence-Based-Guidelines-2023.pdf.
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS consensus workshop group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome (PCOS). Hum Reprod. 2004 Jan;19(1):41-7. doi: 10.1093/humrep/deh098. PMID 14688154
- [Background] Skiba MA, Islam RM, Bell RJ, Davis SR. Understanding variation in prevalence estimates of polycystic ovary syndrome: a systematic review and meta-analysis. Hum Reprod Update. 2018 Nov 1;24(6):694-709. doi: 10.1093/humupd/dmy022. PMID 30059968
- See also: Polycystic Ovary Syndrome and Oxidative Stress-From Bench to Bedside — https://pmc.ncbi.nlm.nih.gov/articles/PMC10531631/